CLINICAL TRIAL: NCT02881905
Title: Peri-Implant Soft Tissue Health and Marginal Bone Loss of Single Implant Mandibular Overdenture Retained by CM LOC Versus Ball Attachment: A Randomised Controlled Trial
Brief Title: PeriImplant Soft Tissue and Marginal Bone Loss of Single Implant Mandibular Overdenture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Ahmed Salah Hamed Sherif, associate lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-8-179
Record Dates: First submitted 2016-08-22; First posted 2016-08-29 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Complete Edentulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ball attachment (Active Comparator): completely edentulous patients having single median mandibular implant to retain mandibular overdenture.the attachment used is the conventional ball attachment
  Interventions: Device: ball attachment
- CM LOC attachment (Experimental): completely edentulous patients having single median mandibular implant to retain mandibular overdenture.the attachment used is the cm loc attachment
  Interventions: Device: cm loc attachment

INTERVENTIONS:
Device: ball attachment — it is attachment part that connects the overdenture to the implant
  Other Names: metallic ball attachment
  Arms: ball attachment
Device: cm loc attachment — It is a new attachment made of peek material
  Arms: CM LOC attachment

SUMMARY:
There is a significant difference between CM LOC and ball attachment, when considering the peri-implant soft tissue health and marginal bone loss. The primary and secondary objectives are to determine if CM LOC attachment improves the peri-implant soft tissue response and decreases the marginal bone loss around implant when compared to conventional ball attachment

DETAILED DESCRIPTION:
Ball attachments are very commonly used because they are solitary, simple, easier to use and less technique sensitive if compared to bar attachments. However, ball attachment require a prosthetic space of 12 mm and could show tremendous wear if implants were mal-aligned. CM LOC attachment is newly introduced into market with very good expectations regarding its properties and effect on the periimplant soft tissue. CM LOC attachment, which combes titanium patrix and resin matrix made from polyetherketoneketone (PEKK), is a very promising material regarding the wear and the prosthesis retention it provides, even with mal-aligned implants. However, the clinical performance of this attachment was not tested yet. Therefore, in this randomized controlled trial it was decided to compare between CM LOC and the commonly used ball attachment regarding the soft tissue health and marginal bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous male or female patients between the ages of 50 to 69.
* No contraindications for implantation.
* Each patient has to perform both a random blood sugar and Glycosylated Hemoglobin analysis. Patients with a Glycosylated hemoglobin test HbA1c up to 8% and a normal blood sugar level (79 to 110) or controlled diabetic patients (90-130 fasting according to American Association of Diabetes) will be included.
* Sufficient bone width (≥ 6 mm) in the anterior region to place an implant. It could be either normally present or achieved by bone plateauing. This will be confirmed by cone beam computed tomographic (CBCT) scans.
* Residual bone height ranging from 11-20 mm with the lowest vertical height in the midline of the mandible not less than 13 mm (Class II or III according to McGarry et al[16] 1999). This will be confirmed by the CBCT.
* Patients seeking to install a single symphyseal implant and for whom new dentures will be constructed.
* Patients, who are dissatisfied with the retention and stability of their technically satisfactory dentures.
* Patients, who already have existing maxillary and mandibular complete dentures, and after examination of the mandibular dentures, it is found that there are technical problems with regard to denture design and/or occlusion; then new maxillary and mandibular dentures will be fabricated
* All patients should have adapted to their dentures for at least six weeks before being included in the trial.
* Patients providing written informed consents to participate in the trial and this will be done before the scheduled date for implant installation.

Exclusion Criteria:

* Patients with a systemic or local contra-indication for implant placement.
* Satisfied patients with the retention of their mandibular denture as well as unsatisfied patients with their maxillary denture.
* Patient with a mandibular denture height less than 6 mm between the base of the denture and the incisal edge of the central incisors (as measured by a caliper) or with 12 mm crown height space as measured by a ruler from the incisal edge till the crest of the ridge. This will be done from a putty index of the diagnostic set up.
* Incompliant and not cooperative patients.
* Patients smoking more than 10 cigarettes per day.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Soft tissue reaction :Presence of mucositis | [from baseline up to 1 year]
  it is a binary outcome that is measured by either its presence or absence

SECONDARY OUTCOMES:
Modified gingival Index | from baseline up to 1 year. score measurement from 0-4 where 0 is no inflammation and 4 is severe inflammation
  0 = absence of inflammation
  1. = mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary
  2. = mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary
  3. = moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary
  4. = severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration. Gingival units as well as the calculation of the index follow the same criteria described in GI
Modified Plaque Index | from baseline upto 1 year. score measurement from 0-3 where 0 denotes no plaque present and 3 denotes abundant plaque
  Modified Plaque Index (mPI) is a dental plaque scale done by Mombelli etal.[13] as follows:
  0 = No plaque
  1. = Separate flecks of plaque at the cervical margin
  2. = Plaque can be seen by naked eye
  3. = Abundance of soft matter. The lower the number the less plaque is present on the tooth
Modified Bleeding Index | from baseline upto 1 year. score from 0-3 where 0 denotes no bleeding and 3 denotes profound bleeding
  Periodontal probe will be passed all around implant cervical margin and bleeding will be scored as follows:
  Score 0: No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant.
  Score 1: Isolated bleeding spots visible.
  Score 2: Blood forms a confluent red line on margin.
  Score 3: Heavy or profuse bleeding.
marginal bone loss | from baseline up to 1 year
  Standardized periapical long cone paralleling technique will be necessary so radiographic template customized for each patient with a holder. Then two reference points will be marked on the implant platform surface and will be joined with a line representing the height zero. then two vertical lines mesial and distal will be drawn to the first bone contact point.

CONTACTS AND LOCATIONS:
Overall Officials: nouran abdelnaby, phd, Study Director — prosthodontic department-faculty of dentistry-cairo university
Locations (1):
- Outpatient Clinic-Prosthodontic Department-Faculty of Dentistry-Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided